CLINICAL TRIAL: NCT04828915
Title: Early Detection of Clinical Deterioration in Patients With COVID-19 Using Machine Learning
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Max-Planck-Institute Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: TEDDI
Record Dates: First submitted 2021-03-24; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-01

CONDITIONS: Covid19
Keywords: Machine learning; Artificial intelligence; Clinical course
MeSH Terms: conditions — COVID-19; Disease Progression | interventions — Machine Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Randomly selection of 80% of the study population. The machine learning algorithm is trained on this dataset
  Interventions: Other: Machine learning
- Validation cohort: Randomly selection of 20% of the study population. The machine learning algorithm which was trained on the basis of the training data cohort is validated on the validation cohort.
  Interventions: Other: Machine based evaluation

INTERVENTIONS:
Other: Machine learning — Machine learning on vital parameters, clinical symptoms and underlying diseases
  Groups: Training cohort
Other: Machine based evaluation — Quantification of the prediction power and identification of the most relevant predictive parameters
  Groups: Validation cohort

SUMMARY:
The aim of this study is to use artificial intelligence in the form of machine learning analysing vital signs as well as symptoms of patients suffering from Covid19 to identify predictors of disease progression and severe course of disease.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >= 18 years
* Detection of SARS-CoV2 within the past 5 days

Exclusion Criteria:

* Inability to measure vital parameters and document symptoms

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with detection of SARS-CoV2
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Probability of Participants for Hospitalisation or Fatal Outcome | Detection of severe acute respiratory syndrome- Corona Virus 2 (SARS-CoV2) to recovery, hospitalisation or fatal outcome up to 5 weeks

SECONDARY OUTCOMES:
Probability of Participants for Intensive Care Unit Admission | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Probability of Participants for Fatal Outcome | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Prediction of persisting health impairment by using standardized questionnaires | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Detection of symptoms, vital parameters and comorbidities predicting clinical course | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Influence of size of training data set | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Influence of viral load on the course of disease/ clinical outcome | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Influence of different virus variants on the course of disease/ clinical outcome | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Influence of SARS-CoV2 vaccination (yes/no) on the course of disease/ clinical outcome | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Evaluation of parameters (symptoms, vital parameters, comorbidities) according to their potential of clinical course predictions | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Probability of Participants for hospitalisation | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks
Influence of different SARS-CoV2 vaccines on the course of disease/ clinical outcome | Detection of SARS-CoV2 to recovery, hospitalisation or fatal outcome up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Schoelkopf, PhD, Study Chair — Max-Planck-Institute, Tuebingen, Germany; Juergen Hetzel, MD, Principal Investigator — University Hospital of Tuebingen, Tuebingen, Germany
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No